CLINICAL TRIAL: NCT06926088
Title: Impact of BMI on CDK4/6 Inhibitors Efficacy and Safety in Advanced Breast Cancer: a Multi-center, Real-world Study
Brief Title: Impact of BMI on CDK4/6 Inhibitors Efficacy and Safety in Advanced Breast Cancer
Acronym: CAMELIA
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CAMELIA
Record Dates: First submitted 2025-03-30; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Advanced Breast Cancer
Keywords: BMI; CDK4/6 Inhibitors
MeSH Terms: interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: BMI < 25.0 kg/m²
  Interventions: Drug: Impact of BMI on CDK4/6 Inhibitors Efficacy and Safety
- Group 2: BMI ≥ 25.0 kg/m²
  Interventions: Drug: Impact of BMI on CDK4/6 Inhibitors Efficacy and Safety

INTERVENTIONS:
Drug: Impact of BMI on CDK4/6 Inhibitors Efficacy and Safety — Patients aged ≥18 years with advanced HR-positive breast cancer who received CDK4/6 inhibitors at six hospitals in China were included in this study.

SUMMARY:
Exploring the Impact of body mass index on the efficacy and safety of CDK4/6 inhibitors combined with endocrine therapy in advanced breast cancer.

DETAILED DESCRIPTION:
Body mass index (BMI) is strongly associated with the development and progression of breast cancer. Despite the widespread use of cyclin-dependent kinase (CDK) 4/6 inhibitors combined with endocrine therapy (ET) in hormone receptor (HR)-positive advanced breast cancer, the effect of BMI on therapeutic outcomes remains poorly understood. Here, we present real-world evidence to substantiate the association between BMI and CDK4/6 inhibitors efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above;
* Women of any menstrual status;
* Histologically confirmed recurrent or metastatic breast cancer, including patients initially diagnosed as stage IV or locally advanced inoperable;
* Patients with histological pathology that is clearly HR-positive/HER2-negative breast cancer, or if there is metastatic pathology, the histological pathology of the metastatic foci shall prevail. (Those with ER intensity >1% cellular nuclear staining)
* Patients have at least 3 more fully documented medical records at the enrolled centre, including at least 1 inpatient record.

Exclusion Criteria:

* CDK4/6 inhibitors as neoadjuvant or adjuvant therapy;
* Significantly missing diagnostic and treatment data from patients' medical records;
* Participation in other clinical trials before and during the data collection period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with advanced HR-positive breast cancer who received CDK4/6 inhibitors at six hospitals in China were included in this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.

SECONDARY OUTCOMES:
Overall Survival (OS) | It is defined as the time from the start of treatment to death for any reason, whichever came first, assessed up to 100 months
  It is defined as the time from the start of treatment to death for any reason.
Objective Response Rate (ORR) | From date of observation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The overall response rate is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set
The Number of Participants Who Experienced Adverse Events | From date of observation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No